CLINICAL TRIAL: NCT00469404
Title: Single Dose Bioequivalence Trial Comparing a Down-Scaled New Analgesic Transdermal Patch Formulation to an Analgesic Reference Patch.
Brief Title: Single Dose Trial Comparing the Plasma Levels of Two Different Analgesic Transdermal Patch Formulations (Protocol ID 297307)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial end was achieved according to the definition in the trial protocol
Sponsor: Grünenthal GmbH (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 297307
Record Dates: First submitted 2007-04-18; First posted 2007-05-04 (Estimated); Last update posted 2007-11-16 (Estimated); Status verified 2007-11

CONDITIONS: Healthy
Keywords: Transdermal patch; Centrally acting analgesic; Plasma level; Healthy volunteers
MeSH Terms: interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to determine whether the plasma levels of two different analgesic transdermal patch formulations lead to same plasma levels of the active ingredient after single dose application.

DETAILED DESCRIPTION:
Main: To demonstrate the bioequivalence between the two transdermal analgesic formulations after single patch application. Pharmacokinetic target parameters are AUC, AUC0-t, and Cmax.

Further: To assess the safety, tolerability, skin tolerability and adhesiveness of the patch applications.

ELIGIBILITY:
Inclusion Criteria:

* Male Caucasian subjects, aged 18-55 years
* BMI between 18 and 30 kg/m2 inclusive, with a lower limit of body weight of 50 kg
* Subjects must be in good health as determined by medical history, physical examination, 12-lead electrocardiogram, vital signs, and clinical laboratory parameters.
* Subjects giving written informed consent to participate within this trial.

Exclusion Criteria:

* Resting pulse rate < 45 or > 100 beats / min
* Resting blood pressure:

systolic blood pressure < 90 and > 160 mmHg, diastolic blood pressure < 40 and > 100 mmHg

* History or presence of orthostatic hypotension
* Positive test of HIV type 1/2 antibodies, HBs antigen, HBc antibodies, HCV antibodies
* Participation in another clinical trial in the last 30 days before starting this trial (i.e., first administration of IMP)
* Positive drug of abuse screening
* Diseases or condition known to interfere with the absorption, distribution, metabolism or excretion of drugs
* Marked repolarisation abnormality (e.g., suspicious or definite congenital long QT syndrome with QT/QTc>500msec or prolonged QTc, i.e.>450msec) or co- medication that is known to influence cardiac repolarisation substantially
* Bronchial asthma
* Definite or suspected history of drug allergy or hypersensitivity
* Subjects who have received any prescribed and non-prescribed systemic or topical medication like analgesics, NSAIDs (except standard dose of a NSAID once a week for the treatment of headache), hypnotics, sedatives, narcotics, neuroleptics or other medications that may lower the seizure threshold, MAO-inhibitors, serotonin-reuptake-inhibitors, tricyclic antidepressants, other centrally acting substances and substances which are known to interact with the drug metabolizing enzymes (e.g., inhibitors or inducers of CYP3A4 or CYP2D6) four weeks prior to the start of the trial (i.e. first administration of IMP). Each case has to be decided upon individually by the investigator after consultation with the Sponsor.
* Evidence of alcohol or drug abuse
* Not able to abstain from consumption of:

Caffeine containing beverages or food (tea, coffee, cola, chocolate, etc.) Quinine containing beverages or food (bitter lemon, tonic water) Grapefruit juice (sweet, sour) Poppy seeds containing beverages or food;

* Blood loss (> 100 mL) due to e.g. blood donation within 3 months before starting this trial (i.e., first administration of IMP)
* History of seizures or at risk (i.e. head trauma, epilepsy in family anamnesis, unclear loss of consciousness)
* Known or suspected of not being able to comply with the trial protocol
* Not able to communicate meaningfully with the investigator and staff
* Smoking of >10 cigarettes/day or equivalent

Trial specific exclusion criteria:

* Subjects not able to abstain from strenuous exercise during the whole course of the trial
* Abnormality (e.g. scar, tattoo) or unhealthy skin at application site according to examination by the investigator
* Existing chronic skin disease or history of skin disease at the application site within the last 4 weeks
* Presence of one of the contraindications as detailed in the current protocol

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2007-05; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Timmer, Dr., Principal Investigator — CRS Clinical Research Services Mannheim
Locations (1):
- Site Mannheim, Mannheim, Germany